CLINICAL TRIAL: NCT02299167
Title: The Minimal Effective Dose of Hyperbaric Spinal Bupivacaine for Successful Reliable Saddle Block for Minor Perianal Surgeries
Brief Title: Minimal Effective Dose of Hyperbaric Spinal Bupivacaine for Saddle Block
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANE-2014-1-23
Record Dates: First submitted 2014-11-19; First posted 2014-11-24 (Estimated); Results first posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-09

CONDITIONS: Perianal Surgery
Keywords: Perianal surgery; hyperbaric bupivacaine; saddle block

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Saddle block (Experimental): The dose of bupivacaine given to each patient was determined by the response of the previously tested patient using a modified Dixon's up-and-down method
  Interventions: Drug: Dixon's up-and-down method

INTERVENTIONS:
Drug: Dixon's up-and-down method — using a modified Dixon's up-and-down method (using 0.5 mg as a step size) (16). The first patient was tested at a dose 1.5 mg bupivacaine, if patient responded with failed block then the next patient received an increment of 0.5mg bupivacaine, if patient responded with successful block, then the next patient received a decrement of 0.5mg bupivacaine. The research continued until we obtained seven crossover midpoints.

SUMMARY:
The optimal anesthetic technique would provide excellent operating conditions, rapid recovery, early discharge, no postoperative side effects, and high patient's satisfaction. In addition to increasing the quality and decreasing the costs of the anesthetic services (1). Selective spinal anesthesia (SSA) -spinal block with minimal effective doses for a specific type of surgery - has become very popular technique) 2(for some orthopedic and gynecological surgeries [3-9].

Saddle anesthesia is a SSA directs a small bolus of hyperbaric local anesthetic, towards S4-S5 and coccygeal nerve roots (11), and is commonly utilized for perianal surgeries (11-14). Hyperbaric bupivacaine has been safely, replaced hyperbaric Lidocaine for saddle block (11, 12).

Although Saddle blocks at different low doses of hyperbaric bupivacaine (1.5- 4 mg) have been used previously for mi¬nor perianal surgeries (11, 13, 14), the optimal effective dose has yet to be determined.

The objective of this study is to determine the minimal effective dose of hyperbaric spinal bupivacaine required to induce a reliable and satisfactory saddle block for perianal surgeries (using a modified Dixon's up-and-down method.

DETAILED DESCRIPTION:
Following approval of the Research and Ethics Committee of the University of Dammam and written informed consent, patients with American Society of Anesthesiologists physical Status I and II, aged 20-55 years, scheduled for outpatient elective perianal surgery in the lithotomy position ( hemorrhoidectomy, fistulectomy), were prospectively enrolled in this study. Patients unwilling to participate, those with contraindications to regional anesthesia, morbid obesity, bleeding disorders, mental health problems or language barriers, taking psychotropic or analgesic medication, or a known history of allergic reactions to amide local anesthetics, were excluded from the study.

Actually, 35 patients were enrolled. However; after they have signed the informed consent; 7 patients were excluded because they have received analgesics in the morning of surgery, and 4 patients refused to receive the saddle block on the operating room. So actually 24 patients out of 35 participants underwent intervention

All patients were fasted for over 6 hours and were premedicated with 0.2 mg/kg oral diazepam 60 min before spinal anesthesia.

In the operating room (OR), an intravenous (IV) 18-20G catheter was placed, and standard monitoring [electrocardiogram (ECG), heart rate (HR), oxygen saturation (SpO2), and noninvasive blood pressure (NIBP)] were started.

Under aseptic conditions, the dural puncture was performed by staff-grade anesthesiologists, using a standard midline approach in the sitting position at the L3-L4 or L4-L5 intervertebral space, using a 25-gauge Whitacre needle with its orifice directed caudally. A predetermined small dose of hyperbaric bupivacaine (Marcaine Spinal Heavy; Astra Zeneca, Lund, Sweden) which was prepared in1 mL tuberculin syringe was injected. All patients remained in the sitting position for 10 min. the patient was asked if he/she perceived any change in motor power.

If not, the patient was allowed to position him/herself without aid for surgery in the lithotomy position. Immediately before surgery, the sacral level of sensory block was tested using a long surgical toothless clamp gently applied radially, starting from the anal orifice, in different diagonal directions.

The motor block was tested by a modified Bromage scale (0 = no motor block, 1 = able to flex the ankle and bend knees, 2 = able to flex ankle, and 3 = full motor block).

A successful block was defined as one that was sufficient to proceed with the surgery without any supplementation (intravenous analgesic, local anesthetic infiltration, or general anesthesia).

The dose of bupivacaine given to each patient was determined by the response of the previously tested patient using a modified Dixon's up-and-down method (using 0.5 mg as a step size) (16).

The first patient was tested at a dose 1.5 mg bupivacaine, if the patient responded with a failed block then the next patient received an increment of 0.5 mg bupivacaine, if the patient responded with a successful block, then the next patient received a decrement of 0.5 mg bupivacaine.

The research continued until the investigators obtained seven crossover midpoints. The initial starting dose of 1.5 mg hyperbaric bupivacaine of the first patient was selected from the findings of Wassef R et al. who demonstrated adequate anesthesia for short perianal surgery with the use of 1.5 mg spinal hyperbaric bupivacaine.

Bupivacaine was prepared immediately before injection by an independent anesthesiologist and was administered by a second anesthesiologist. Block assessment and clinical follow-up of the patients was also performed by a third anesthesiologist.

The following data were recorded; Patient demographics, duration of anesthesia and surgery, level of sensory and motor block immediately before surgery, at the end of the surgery, and every 30 minutes until resolution of the block. NIBP and HR were documented every 5 minutes in the OR and PACU. Also Times to ambulation, first voiding time, and time to home discharge were recorded. Patient's and surgeon's satisfaction were evaluated with a 4-point score (0=poor, 1=good, 2=very good, 3= excellent). Patients were followed by phone call to note down any possible postoperative complication (postdural puncture headache, TNS or backache) at day 1 postoperatively and 10 days later. The time of the dural puncture was used as the primary starting point of assessment.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical Status I and II patients.
* Scheduled for outpatient elective perianal surgery.

Exclusion Criteria:

* Patients unwilling to participate.
* Contraindications to regional anesthesia.
* Morbid obesity.
* Bleeding disorders.
* Mental health problems.
* Language barrier.
* Taking psychotropic or analgesic medication.
* History of allergic reactions to amide local anesthetics.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roshdi Al Metwalli, MD, Principal Investigator — Associate Professor at Anesthesiology Dept

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four independent anesthetists were assigned for the study from January 2014.one to select patients in the anesthesia clinic, the 2nd to prepare the studied drug in the OR, the 3rd one to inject the drug and the 4th one was to collect the data
Pre-assignment Details: 35 patients were enrolled However; after they have signed the consent. 7 patients were excluded because they have received analgesics in the morning of surgery. and 4 patients refused the saddle block in the operating room. So actually 24 patients out of 35 participants underwent intervention. That has been already specified in the protocol
Groups:
- Single Group Study / Saddle Block: The dose of bupivacaine given to each patient was determined by the response of the previously tested patient using a modified Dixon's up-and-down method
  Dixon's up-and-down method: using a modified Dixon's up-and-down method (using 0.5 mg as a step size) (16). The first patient was tested at a dose 1.5 mg bupivacaine, if patient responded with failed block then the next patient received an increment of 0.5mg bupivacaine, if patient responded with successful block, then the next patient received a decrement of 0.5mg bupivacaine. The research continued until we obtained seven crossover midpoints.
Period: Overall Study
Arm/Group | Single Group Study / Saddle Block
Started | 35
Dural Puncture (Dural puncture to inject the study drug) | 24
Success Rate (10 min after Dural puncture (to test the success of the block)) | 24
Adverse Effects (24 after surgery to record any complication) | 24
Completed | 24
Not Completed | 11
Not completed — patients were excluded from the study | 11

BASELINE CHARACTERISTICS:
Population: 11 patients have been excluded from the study. The remaining 24 participants completed the study
Arm/Group | Saddle Block
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants] — 11 patients have been excluded from study. The remaining 24 participants completed the study.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 24
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.71 (10.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 24
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Saudi Arabia | 24

OUTCOME MEASURES:

1. Primary Outcome: Minimal Effective Dose of Hyperbaric Bupivacaine
Description: the minimal effective dose of hyperbaric bupivacaine using a modified Dixon's up-and-down method (using 0.5 mg as a step size) (16). The first patient was tested at a dose 1.5 mg bupivacaine, if patient responded with failed block then the next patient received an increment of 0.5mg bupivacaine, if patient responded with successful block, then the next patient received a decrement of 0.5mg bupivacaine. The research continued until we obtained seven crossover midpoints.
Time Frame: 10 min after dural puncture
Measure: Mean (95% Confidence Interval); unit: milligrams
Arm/Group | Single Group Study / Saddle Block
Number analyzed (Participants) | 24
milligrams | 1.9 [1.7 to 2.1]
Statistical Analysis 1: Comparison: Single Group Study / Saddle Block; Descriptive statistics were considered to calculate the mathematic mean (SD) of demographic, surgical, and other postoperative continuous data and to calculate the median (range) of sensory and motor block levels, as well as the degree of patient and surgeon satisfaction; Test type: Other — The ED50% of spinal bupivacaine was estimated using a modified Dixon's up-and-down method; Mean (95% CI) of effective dose in 90% ( = 1.9, 95% CI 2-sided [1.7 to 2.1] — The ED50% of spinal bupivacaine was estimated using a modified Dixon's up-and-down method

2. Secondary Outcome: Sacral Level of Sensory Block
Description: The level of sensory block was tested using a long surgical toothless clamp gently applied radially, starting from the anal orifice, in different diagonal directions
Time Frame: every 30 min until complete regression of the block (approximately 90 min)
Population: * Immediately before surgery S4 (S3-S4)
  * At conclusion of surgery S4 (S3-S4)
  * Maximum blocked dermatome S4 (S3-S4)
Measure: Median (Full Range); unit: Sacral level of sensory block
Arm/Group | Single Group Study / Saddle Block
Number analyzed (Participants) | 12
Sacral level of sensory block
  Maximum blocked dermatome | 4 [3 to 4]
  At conclusion of surgery | 4 [3 to 4]
  Immediately before surgery | 4 [3 to 4]

3. Secondary Outcome: Motor Block Score as Assessed Using the Bromage Scale
Description: The motor block was tested by a modified Bromage scale (0 = no motor block, 1 = able to flex the ankle and bend knees, 2 = able to flex ankle, and 3 = full motor block). A successful block was defined as one that was sufficient to proceed with the surgery without any supplementation (intravenous analgesic, local anesthetic infiltration, or general anesthesia).
Time Frame: every 30 min until Time to ambulation (approximately 2 hours)
Population: The block characteristics for patients with successful block (12 patients)
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Single Group Study / Saddle Block
Number analyzed (Participants) | 12
score on a scale
  Immediately before surgery | 0 [0 to 0]
  At conclusion of surgery 0 Aided patient positioni | 0 [0 to 0]

4. Secondary Outcome: Patient's Satisfactions
Description: Patient's satisfactions were evaluated with a 4-point satisfaction score (0=poor satisfaction, 1=good satisfaction 2=very good satisfaction, 3= excellent satisfaction
Time Frame: 24 hours after surgery
Population: All patient with successful block were satisfied
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Single Group Study / Saddle Block
Number analyzed (Participants) | 12
score on a scale | 3 [2 to 3]

5. Secondary Outcome: Surgeon's Satisfactions
Description: Surgeon's satisfactions were evaluated with a 4-point satisfaction score (0=poor satisfaction, 1=good satisfaction 2=very good satisfaction, 3= excellent satisfaction
Time Frame: 24 hours after procedure
Population: All surgeon who operated on the patient with successful block (12 patients ) were satisfied
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Single Group Study / Saddle Block
Number analyzed (Participants) | 12
score on a scale | 3 [2 to 3]

ADVERSE EVENTS:
Time Frame: 24 hours
Description: Postoperative complications
  PDPH 0 (0-0) Urinary retention 0 (0-0) backache 0 (0-0)
Groups:
- Single Group Study / Saddle Block: The dose of bupivacaine given to each patient was determined by the response of the previously tested patient using a modified Dixon's up-and-down method (using 0.5 mg as a step size) (16). The first patient was tested at a dose 1.5 mg bupivacaine, if the patient responded with a failed block then the next patient received an increment of 0.5mg bupivacaine, if the patient responded with a successful block, then the next patient received a decrement of 0.5mg bupivacaine. The research continued until we obtained seven crossover midpoints.
Arm/Group | Single Group Study / Saddle Block
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes